CLINICAL TRIAL: NCT07169461
Title: Effectiveness of Low Level Light Therapy and Intense Pulse Light on Mite Count as Adjuntive Therapies in Demodex Blepharitis Using Artificial Intelligent Program (Ai-Demodex): A Factorial Randomized Sham-Controlled Trial
Brief Title: Effectiveness of Low Level Light Therapy and Intense Pulse Light on Mite Count as Adjuntive Therapies in Demodex Blepharitis Using Artificial Intelligent Program (Ai-Demodex)
Acronym: Ai-Demodex
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Other
Other Study IDs: 40567
Record Dates: First submitted 2025-03-11; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-01

CONDITIONS: Demodex Blepharitis; Meibomian Gland Dysfunction (MGD)
Keywords: Demodex blepharitis; MGD; Meibomian gland dysfunction; Low level light therapy; LLLT; Intense Pulse Light Therapy; IPL; Demodex mite count; Ocular surface parameters; Demodex mite eradication; Ai in demodex; Ai in MGD
MeSH Terms: conditions — Meibomian Gland Dysfunction | interventions — Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- ShamLLLT plus ShamIPL (Sham Comparator): ShamLLLT : the MY MASK-E (Espansione Marketing S.p.A., Bologna, Italy) - No eye shields, applying a power off special mask for 15 minutes , once a week for 4 weeks ShamIPL : the Eye-light device (Espansione Marketing S.p.A., Bologna, Italy) - Protective eye shields, 5 time for each eye with flashes of light off , but flashes sound on.
  with Mechanical with pharmacological treatment : Warm compression 15 minutes + Lid hygiene + 1% TTO for 90 days
  1%TTO : OCuSOFT Oust Demodex Eyelid Cleanser Foam Bottle 50ml (OCuSOFT, Richmond, TX) is the only commercially available medication in Thailand that contains 1% tea tree oil.
  Interventions: Procedure: Mechanical with pharmacological treatment; Device: ShamIPL; Device: ShamLLLT
- LLLT plus ShamIPL (Experimental): LLLT : The blue MY MASK-E (Espansione Marketing S.p.A., Bologna, Italy) (Thai FDA No 66-2-2-2-0012685)
  * No eye shields
  * Applying a special mask for 15 minutes, once a week for 4 weeks
  ShamIPL : the Eye-light device (Espansione Marketing S.p.A., Bologna, Italy) - Protective eye shields, 5 time for each eye with flashes of light off.but flashes sound on.
  with Mechanical with pharmacological treatment : Warm compression 15 minutes + Lid hygiene + 1% TTO 2 times per day for 90 days
  1%TTO : OCuSOFT Oust Demodex Eyelid Cleanser Foam Bottle 50ml (OCuSOFT, Richmond, TX) is the only commercially available medication in Thailand that contains 1% tea tree oil.
  Interventions: Device: The blue MY MASK-E; Procedure: Mechanical with pharmacological treatment; Device: ShamIPL
- IPL plus ShamLLLT (Experimental): IPL : The Eye-light device (Espansione Marketing S.p.A., Bologna, Italy,waveleggths 1,200-1,500 nm, Delivery system 12cm2) (Thai FDA No 66-2-2-2-0012685) :
  * Protective eye shields
  * 5 flashes of light were applied for each eye (3 along the inferior orbital rim, 1 at the lateral canthus, and 1 applied horizontally along the inferior orbital rim)
  * Therapeutic energy level (10-16 joules/ cm2) based on the degree of skin pigmentation.
  ShamLLLT : the MY MASK-E (Espansione Marketing S.p.A., Bologna, Italy) - No eye shields, applying a power off special mask for 15 minutes , once a week for 4 weeks
  with Mechanical with pharmacological treatment : Warm compression 15 minutes + Lid hygiene + 1% TTO 2 times per day for 90 days
  1%TTO : OCuSOFT Oust Demodex Eyelid Cleanser Foam Bottle 50ml (OCuSOFT, Richmond, TX) is the only commercially available medication in Thailand that contains 1% tea tree oil.
  Interventions: Device: IPL; Procedure: Mechanical with pharmacological treatment; Device: ShamLLLT
- LLLT plus IPL (Experimental): IPL : The Eye-light device (Espansione Marketing S.p.A., Bologna, Italy,waveleggths 1,200-1,500 nm, Delivery system 12cm2) (Thai FDA No 66-2-2-2-0012685) :
  * Protective eye shields
  * 5 flashes of light were applied for each eye (3 along the inferior orbital rim, 1 at the lateral canthus, and 1 applied horizontally along the inferior orbital rim)
  * Therapeutic energy level (10-16 joules/ cm2) based on the degree of skin pigmentation.
  LLLT : The blue MY MASK-E (Espansione Marketing S.p.A., Bologna, Italy) (Thai FDA No 66-2-2-2-0012685)
  * No eye shields
  * Applying a special mask for 15 minutes, once a week for 4 weeks with Mechanical with pharmacological treatment : Warm compression 15 minutes + Lid hygiene + 1% TTO 2 times per days for 90 days 1%TTO : OCuSOFT Oust Demodex Eyelid Cleanser Foam Bottle 50ml (OCuSOFT, Richmond, TX) is the only commercially available medication in Thailand that contains 1% tea tree oil.
  Interventions: Device: The blue MY MASK-E; Device: IPL; Procedure: Mechanical with pharmacological treatment

INTERVENTIONS:
Device: The blue MY MASK-E — Device-Specific Protocol Blue MyMask® LLLT (Espansione): Emits monochromatic photobiomodulation therapy at 633 nm, distinct from conventional red or near-infrared LLLT used in other studies.
  Espansione IPL: Uses a patented Optimal Power Energy (OPE®) system with a polychromatic spectrum of 590-1200 nm, allowing sub-threshold energy pulses for selective thermal effects on abnormal telangiectasia and Demodex-related inflammation.
  Arms: LLLT plus IPL; LLLT plus ShamIPL
Device: IPL — IPL : The Eye-light device (Espansione Marketing S.p.A., Bologna, Italy,waveleggths 1,200-1,500 nm, Delivery system 12cm2) (Thai FDA No 66-2-2-2-0012685) :
  * Protective eye shields
  * 5 flashes of light were applied for each eye (3 along the inferior orbital rim, 1 at the lateral canthus, and 1 applied horizontally along the inferior orbital rim)
  * Therapeutic energy level (10-16 joules/ cm2) based on the degree of skin pigmentation.
  Arms: IPL plus ShamLLLT; LLLT plus IPL
Procedure: Mechanical with pharmacological treatment — Mechanical with pharmacological treatment : Warm compression 15 minutes + Lid hygiene + 1% TTO 2 times per day for 90 days
  1%TTO : OCuSOFT Oust Demodex Eyelid Cleanser Foam Bottle 50ml (OCuSOFT, Richmond, TX) is the only commercially available medication in Thailand that contains 1% tea tree oil.
Device: ShamIPL — the Eye-light device (Espansione Marketing S.p.A., Bologna, Italy) - Protective eye shields, 5 time for each eye with flashes of light off , but flashes sound on.
  Arms: LLLT plus ShamIPL; ShamLLLT plus ShamIPL
Device: ShamLLLT — the MY MASK-E (Espansione Marketing S.p.A., Bologna, Italy) - No eye shields, applying a power off special mask for 15 minutes but light on , once a week for 4 weeks
  Arms: IPL plus ShamLLLT; ShamLLLT plus ShamIPL

SUMMARY:
Primary Objective:

To evaluate the efficacy of LLLT, IPL, and IPL + LLLT in re ducing demodex count in patients with Demodex Blepharitis.

Secondary Objectives:

To evaluate the efficacy of LLLT, IPL, and IPL + LLLT in improving ocular surface parameters in Demodex Blepharitis.

Sample Size:

88 participant ( 22 participants per group x 4 groups)

Study Design:

2x2 Factorial randomized trial.

Methodology:

The study is composed of 4 groups including 1) control 2) Blue light LLT alone 3) IPL alon e, 4) Blue light LLLT with IPL , and .

Both LLLT and IPL will treat weekly for 4 sessions All participants will be instructed to perform warm compression and lid scrub. The outcomes include demodex count, meibum grading and ocular surface parameter were evaluated at 1 and 3 months post treatment.

ELIGIBILITY:
Inclusion Criteria:

1. All patients who received a definite diagnosis of demodex blepharitis based on cylindrical dandruff at the base of the lashes and the presence of at least one alive demodex mites on eyelid margin by microscopy
2. Age >18 years.
3. Patients who can understand and follow the study instructions and can adhere to the scheduled follow-up plan.

Exclusion Criteria:

1. Patients who received previous treatment IPL or LLLT
2. Poor compliance with eyelid scrubbing using tea tree oil (TTO)
3. Dead demodex mite on lash.
4. Contraindication of IPL: Skin Fitzpatrick scale V/VI, patients with pigmented lesions on the treatment area (Eyelid, Cheek).
5. Pregnancy or breastfeeding.
6. Active Skin disease: facial skin cancer, graft-versus-host disease, systemic lupus erythaematosus
7. Active eye infection: recurrent herpes simplex
8. Other lid disease ocular trauma, ocular deformity scar, exophthalmos, eyelid insufficiency
9. Patients with pigmented lesion on area of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Mean of Demodex Count in 30 days after treatment | 30 days after end of treatment. (8th week)
  The number of Demodex mites per eyelash on a total of 4 collarettes lashes epilation (2 from upper eyelid ,2 from lower eyelid and identification by anatomical imaginary line of nasal and temporal limbus) per right eye in 30 days after end of treatment.
  (8th week)

SECONDARY OUTCOMES:
Mean of Demodex Count in 90 days after treatment | 90 days after end of treatment. (16th week)
  Mean of Demodex Count in 90 days after treatment per right eye in 90 days after end of treatment.(16th week)
MGD staging (Severity) | Day 0, 8th week,16th week
  OSDI questionnaire used to evaluate ocular dry eye symptoms. Meibum Quality. Meibum Expressibility. Telangiectasia grading: 0-3
Surface Staining: NEI Grading System. | Day 0 , 8th week ,16th week
Lipid Layer Thickness by LIPIVIEW | Day 0 , 8th week , 16th week
Noninvasive break-up time (NIBUT) | Day 0, 8th week,16th week
Tear meniscus height (TMH) | Day 0 , 8th week ,16th week
% Meibomian Gland Loss (MGL) | Day 0 , 8th week ,16th week

CONTACTS AND LOCATIONS:
Overall Officials: Vannarut Satitpitakul, MD, Principal Investigator — Department of ophthalmology, Faculty of Medicine
Locations (1):
- Chulalongkorn University, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT07169461/Prot_SAP_000.pdf
  • Informed Consent Form (2024-12-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT07169461/ICF_001.pdf